CLINICAL TRIAL: NCT04265885
Title: Gender Dysphoria and Transition: Testimony From Transgender People
Brief Title: Gender Dysphoria and Transition
Acronym: DyGePeT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI033
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collection of testimonies from transgender people — guided interview

SUMMARY:
Persons with gender dysphoria present the difficulties of access to health care. Little time is devoted to education of health professionals about the care of transgender persons. According to the proposal of the French Ministry of Social Affairs and Health there is a need to increase knowledge in this area and to improve the care of transgender people including prevention and screening.

Similarly, little is known about social and medical needs of the transgender population.

This project proposes to illustrate gender dysphoria through testimonies of transgender people with the aim to increase the investigator's understanding aout the needs and the desires of this population and to describe the process of medical and social transition.

ELIGIBILITY:
Inclusion Criteria:

* Person affiliated to a social security system
* Person having received complete information on the organisation of the research and having signed the informed consent
* Person having carried out a prior clinical examination adapted to the research
* Age> 18 years
* Diagnosis of gender incongruence (dysphoria) according to the international classification of diseases, revision 11

Exclusion Criteria:

* Severe, uncontrolled psychiatric or somatic illness
* Substance and alcohol addiction
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participation to the study will be offered consecutively to adult subjects with gender dysphoria followed in the department of endocrinology, diabetology and nutrition of the University Hospital of Nancy.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Illustrate the real-life experiences of transgender people | 4 months

IPD SHARING:
Plan to Share IPD: Undecided